CLINICAL TRIAL: NCT01139437
Title: A Phase I Study of the Safety and Immunogenicity of the Recombinant Live-Attenuated Human Parainfluenza Type 2 Virus Vaccine, rHPIV2 15C/948L/Δ1724 Lot PIV2#109C, Delivered as Nose Drops to Adults 18 to 49 Years of Age, HPIV2-Seropositive Children 15 to 59 Months of Age, and HPIV2-Seronegative Infants and Children 6 to 59 Months of Age
Brief Title: Safety of a Live Attenuated Human Parainfluenza Virus Type 2 (HPIV2) Vaccine for Adults, Children, and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIR 258
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Human Parainfluenza Virus 2
Keywords: Vaccine; HPIV2; Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Adults (Experimental): Adults ages 18 to 49 years of age. Open label.
  Interventions: Biological: Standard Dose HPIV2 Vaccine
- Seropositive children - vaccine (Experimental): Children ages 15 to 59 months of age who already have HPIV2 antibodies receiving the HPIV2 vaccine.
  Interventions: Biological: Standard Dose HPIV2 Vaccine
- Seronegative infants and children - low dose vaccine (Experimental): Infants and children ages 6 to 59 months of age who do not have HPIV2 antibodies receiving a low dose of the HPIV2 vaccine.
  Interventions: Biological: Low dose HPIV2 vaccine
- Seronegative infants and children - standard dose vaccine (Experimental): Infants and children ages 6 to 59 months of age who do not have HPIV2 antibodies receiving a standard dose of the HPIV2 vaccine.
  Interventions: Biological: Standard Dose HPIV2 Vaccine
- Seropositive children - placebo (Placebo Comparator): Children ages 15 to 59 months of age who already have HPIV2 antibodies receiving a placebo.
  Interventions: Other: Placebo
- Seronegative infants and children - low dose placebo (Placebo Comparator): Infants and children ages 6 to 59 months of age who do not have HPIV2 antibodies receiving a low dose of placebo.
  Interventions: Other: Placebo
- Seronegative infants and children - standard dose placebo (Placebo Comparator): Infants and children ages 6 to 59 months of age who do not have HPIV2 antibodies receiving a standard dose of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Standard Dose HPIV2 Vaccine — 10^6 tissue culture infectious dose 50% (TCID50) administered intranasally in a single dose
  Arms: Adults; Seronegative infants and children - standard dose vaccine; Seropositive children - vaccine
Biological: Low dose HPIV2 vaccine — 10^5 TCID50 administered in a single dose
  Arms: Seronegative infants and children - low dose vaccine
Other: Placebo — Matched placebo
  Arms: Seronegative infants and children - low dose placebo; Seronegative infants and children - standard dose placebo; Seropositive children - placebo

SUMMARY:
Human parainfluenza virus type 2 (HPIV2) can result in severe respiratory illness in infants and young children. This study will test the safety of and immune response to an HPIV2 vaccine aimed at infants and children.

DETAILED DESCRIPTION:
HPIV2 is a virus that can cause severe respiratory illnesses, such as pneumonia and bronchiolitis, in infants and young children. Approximately 3% of all hospitalizations for respiratory tract diseases among infants and children are the result of HPIV2. Efforts to develop a vaccine for HPIV2 have focused on a live attenuated intranasally administered vaccine, a type of vaccine that uses a live virus that has been modified to make it weaker and easier for the immune system to get rid of. This approach is useful for several reasons: it activates two of the body's natural defenses, the antibody-mediated and the cell-mediated responses; it is immunogenic in infants who still have maternal antibodies; and it induces a mucosal immune response. This study will test the safety and immunogenicity of an HPIV2 vaccine in adults, children, and then infants.

This study will have four groups and will proceed in a step-wise fashion. The first group will consist only of adults receiving the HPIV2 vaccine. If it is deemed safe after that, children from ages 15 to 59 months who already have HPIV2 antibodies will be randomly assigned to receive either the vaccine or a placebo. The third group includes infants and children from 6 to 59 months old who do not have HPIV2 antibodies and will be randomly assigned either a lower dose of the vaccine or a placebo. The fourth group also includes infants and children from 6 to 59 months old who do not have HPIV2 antibodies and will be randomly assigned a standard dose vaccine or placebo. The vaccine will be administered as a nose drop in a single dose for all groups.

Assessments for the first two groups will take place over the 11 days following administration of the vaccine and at a 28-day follow-up. The third and fourth groups will include 22 days of assessments after vaccination, one assessment between Days 23 and 26, and assessments on Days 27, 28, 29, and 56. Measures will include a clinical assessment, a nasal wash, a phone report, and taking a temperature. Measurement of serum HPIV2 antibodies will take place at baseline and after 28 (for groups one and two) or 56 (for groups three and four) days.

ELIGIBILITY:
Inclusion Criteria for Adults:

* 18 to 49 years old
* In good health, measured by lack of significant medical illness, physical examination findings, or significant laboratory abnormalities of urinalysis, complete blood count (CBC), ALT, or creatinine, as determined by the investigator

Exclusion Criteria for Adults:

* Pregnancy
* Breastfeeding
* Females of childbearing potential who are unwilling to practice effective birth control
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, or laboratory studies, including urinalysis
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the participant to understand and cooperate with the study protocol
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the study or would render the participant unable to comply with the protocol
* Has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* History of a severe allergic reaction or anaphylaxis
* History of splenectomy
* Diagnosis of asthma within the past 2 years
* Positive enzyme-linked immunoassay (ELISA) and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory immunoblot tests for hepatitis C virus (HCV)
* Positive ELISA hepatitis B surface antigen (HBsAg) test
* Abnormal urinalysis or urine dip
* Known immunodeficiency syndrome
* Current use of nasal or systemic steroid medications
* Receipt of blood products (including immunoglobulin) within the past 3 months
* Current smoker unwilling to stop smoking for the duration of the study
* Participation in another investigational vaccine or drug study within 30 days of receiving the investigational vaccine
* Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks or immune globulin within the last 3 months prior to receiving the investigational vaccine
* Previous immunization with an HPIV2 vaccine
* Known hypersensitivity to any vaccine component
* Professional or personal responsibilities involve caring for children less than 59 months of age or for immunosuppressed individuals
* Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Body mass Index (BMI) greater than 35

Inclusion Criteria for Seropositive Children:

* Children 15 to 59 months of age
* Parent or guardian understands and signs the informed consent
* Seropositive for HPIV2, as defined by serum hemagglutinin inhibition (HAI) antibody titer in ratio greater than 1:8
* History has been reviewed and participant has undergone a physical examination indicating good health
* Participant is expected to be available for the duration of the study

Exclusion Criteria for Seropositive Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy, including systemic corticosteroids or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an HPIV2 vaccine
* Current use of nasal or systemic steroid medications
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease. Participants with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. Participants who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 6 months of age
* Attends day care with infants less than 6 months of age or immunosuppressed individuals, and parent or guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable
* Participation in another investigational vaccine or drug trial within 30 days of receiving the investigational vaccine, or while this study is ongoing

Inclusion Criteria for Seronegative Infants and Children:

* Children and infants 6 to 59 months of age
* Parents or guardians can understand and sign the informed consent
* Seronegative for HPIV2 antibody, as defined by serum antibody titer HAI ratio less than or equal to 1:8, as determined within 28 days prior to inoculation
* History has been reviewed and subject has undergone a physical examination indicating good health
* Participant is expected to be available for the duration of the study

Exclusion Criteria for Seronegative Infants and Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy, including systemic corticosteroids or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an HPIV2 vaccine
* Current use of nasal or systemic steroid medications
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease. Participants with clinically insignificant cardiac abnormalities requiring no treatment and those who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may be enrolled.
* Member of a household that includes an immunocompromised individual or infant less than 6 months of age
* Attends day care with infants less than 6 months of age or immunosuppressed individuals, and parent or guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.
* Participation in another investigational vaccine or drug trial within 28 days of receiving the investigational vaccine, or while this study is ongoing

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety, as determined by frequency of adverse events | Measured at baseline, for 11 days after vaccination, and at 1 month follow-up
Immunogenicity, as determined by ability to cause an immunological reaction and amount of antibody induced by the vaccine | Measured at baseline and at 1 month
Infectivity, as determined by amount of vaccine shed by each recipient | Measured at baseline, for 11 days after vaccination, and at 1 month follow-up

SECONDARY OUTCOMES:
Phenotypic stability of the vaccine virus shed | Measured at baseline and at 1 month
Number of vaccinated infants and children infected with HPIV2 | Measured at baseline, for 11 days after vaccination, and at 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins University, Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Murphy BR, Prince GA, Collins PL, Van Wyke Coelingh K, Olmsted RA, Spriggs MK, Parrott RH, Kim HW, Brandt CD, Chanock RM. Current approaches to the development of vaccines effective against parainfluenza and respiratory syncytial viruses. Virus Res. 1988 Aug;11(1):1-15. doi: 10.1016/0168-1702(88)90063-9. PMID 2845680
- [Background] Nolan SM, Skiadopoulos MH, Bradley K, Kim OS, Bier S, Amaro-Carambot E, Surman SR, Davis S, St Claire M, Elkins R, Collins PL, Murphy BR, Schaap-Nutt A. Recombinant human parainfluenza virus type 2 vaccine candidates containing a 3' genomic promoter mutation and L polymerase mutations are attenuated and protective in non-human primates. Vaccine. 2007 Aug 21;25(34):6409-22. doi: 10.1016/j.vaccine.2007.06.028. Epub 2007 Jul 3. PMID 17658669